CLINICAL TRIAL: NCT00772577
Title: An 8-Week Prospective, Multicenter, Randomized, Double-Blind, Active Control, Parallel Group Study to Evaluate the Efficacy and Safety of Aliskiren HCTZ vs Ramipril in Obese Patients (BMI ≥ 30) With Stage 2 Hypertension
Brief Title: Study of the Efficacy and Safety of Aliskiren HCTZ vs Ramipril in Obese Patients (BMI ≥ 30) With Stage 2 Hypertension
Acronym: ATTAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100AUS07
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2011-03-02 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Hypertension, Obese, aliskiren, hydrochlorothiazide, systolic blood pressure, diastolic blood pressure, ramipril, stage 2
MeSH Terms: conditions — Hypertension; Obesity | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aliskiren Hydrochlorothiazide(HCTZ)
  Interventions: Drug: Aliskiren Hydrochlorothiazide
- 2 (Active Comparator): Ramipril
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Aliskiren Hydrochlorothiazide — Aliskiren HCTZ 150/12.5 mg: 1 week; Aliskiren HCTZ 300/25 mg: 7 weeks
  Arms: 1
Drug: Ramipril — Ramipril 5mg: 1 week; Ramipril 10 mg: 7 weeks
  Arms: 2

SUMMARY:
Study to Evaluate the Efficacy and Safety of Aliskiren Hydrochlorothiazide (HCTZ) vs Ramipril in Obese patients (BMI ≥ 30) with Stage 2 Hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible and able to participate in the study, and who give written informed consent before any assessment is performed.
* Male or female outpatients, 18 years of age and older.
* Patients with Stage 2 hypertension. Patients must have a MSSBP ≥ 160 mmHg and < 200 mmHg at Study Visit 5 (randomization).
* Patients must have a BMI ≥ 30 kg/m2 but ≤ 45 kg/m2.

Exclusion Criteria:

* Office blood pressure measured by cuff (MSDBP ≥ 110 mmHg and/or MSSBP ≥ 200 mmHg) at any visit.
* Use of other investigational drugs within 30 days of enrollment, or 5 half-lives, which ever is longer.
* Use of aliskiren and/or a fixed dose combination of aliskiren HCTZ or participation in a clinical trial that had aliskiren and/or aliskiren HCTZ as treatment within 30 days of Visit 1.
* History of hypersensitivity to any of the study drugs or to drugs belonging to the same therapeutic class (ACE inhibitors or renin inhibitors) as the study drugs.
* History or evidence of a secondary form of hypertension.
* Refractory hypertension, defined as, unresponsive to triple drug therapy at the maximum dose of each drug, one of which must be a diuretic, and not at blood pressure goal (140/90 mmHg). Therapy with a fixed dose combination of two active substances represent two drugs.
* Patients on 4 or more antihypertensive medications.
* Long QT syndrome or QTc > 450 msec for males and > 470 msec for females at screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (6):
- United States (6):
  - Investigative Site, Beverly Hills, California
  - Investigative Site, Santa Ana, California
  - Investigative Site, Conyers, Georgia
  - Investigative Site, Lexington, Kentucky
  - Investigative Site, Columbia, South Carolina
  - Investigative Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren HCTZ: Aliskiren HCTZ 150/12.5 mg: 1 week; Aliskiren HCTZ 300/25 mg: 7 weeks
Period: Overall Study
Arm/Group | Aliskiren HCTZ | Ramipril
Started | 193 | 193
Completed | 170 | 170
Not Completed | 23 | 23
Not completed — Adverse Event | 6 | 3
Not completed — Abnormal laboratory values | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 8
Not completed — Patient withdrew consent | 8 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Administrative problems | 2 | 1
Not completed — Protocol Deviation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren HCTZ | Ramipril | Total
Number analyzed (Participants) | 193 | 193 | 386
Age Continuous [Mean (Standard Deviation); unit: years] | 55.4 (11.15) | 54.4 (10.90) | 54.9 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 99 | 206
  Male | 86 | 94 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP)
Description: To assess the change in mean sitting systolic blood pressure (MSSBP) after 8 weeks of treatment with aliskiren HCTZ (150/12.5 mg, 300/25 mg) versus ramipril (5 mg, 10 mg).
Time Frame: Baseline to week 8
Population: Intent-to-treat population (consisted of all patients who received at least one dose of study medication and had at least one valid post baseline assessment of primary efficacy variable). Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren HCTZ | Ramipril
Number analyzed (Participants) | 190 | 190
mm Hg
  Baseline | 167.0 (7.05) | 168.2 (7.86)
  Week 8 | 138.9 (16.56) | 151.6 (17.44)
  Change from baseline to week 8 | -28.1 (15.54) | -16.6 (14.76)

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP)
Description: To evaluate the difference in mean sitting diastolic blood pressure (MSDBP) after 8 weeks of treatment with aliskiren HCTZ (150/12.5 mg, 300/25 mg) versus ramipril (5 mg, 10 mg).
Time Frame: Baseline to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren HCTZ | Ramipril
Number analyzed (Participants) | 190 | 190
mm Hg
  Baseline | 94.3 (8.41) | 96.3 (8.48)
  Week 8 | 84.2 (9.80) | 92.7 (11.07)
  Change from baseline to week 8 | -10.1 (9.04) | -3.6 (9.48)

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control During 8 Weeks
Description: The percentage of patients achieving the Blood Pressure control (defined as patients achieving a MSSBP < 140 mm Hg and MSDBP < 90 mm Hg) during 8 weeks of treatment with aliskiren HCTZ (150/12.5 mg, 300/25 mg) versus ramipril (5 mg, 10 mg). Data presented are cumulative. Cumulative refers to achieving blood pressure control before or at the 8 week visit. If achieving blood pressure control occurred more than once, only the first occurrence was counted.
Time Frame: 8 weeks
Population: Intent-to-treat population (consisted of all patients who received at least one dose of study medication and had at least one valid post baseline assessment of primary efficacy variable).
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren HCTZ | Ramipril
Number analyzed (Participants) | 190 | 190
Percentage of patients | 63.7 | 30.0

4. Secondary Outcome: Percentage of Responders (MSSBP < 140 mmHg or ≥ 20 mmHg Decrease From Baseline in MSSBP)
Description: To compare the percentage of responders (as defined by patients with MSSBP < 140 mm Hg or a decrease from baseline ≥ 20 mm Hg) during 8 weeks of treatment with aliskiren HCTZ (150/12.5 mg, 300/25 mg) versus ramipril (5 mg, 10 mg). Data presented are cumulative. Cumulative refers to achieving the response before or at the 8 week visit. If response occurred more than once, only the first occurrence was counted.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of patients
Arm/Group | Aliskiren HCTZ | Ramipril
Number analyzed (Participants) | 190 | 190
Percentage of patients | 87.9 | 63.2

5. Secondary Outcome: Change From Baseline in Mean Sitting Pulse Pressure (MSPP)
Description: To compare the change in mean sitting pulse pressure (MSPP) after 8 weeks of treatment with aliskiren HCTZ (150/12.5 mg, 300/25 mg) versus ramipril (5 mg, 10 mg).
Time Frame: Baseline to week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Aliskiren HCTZ | Ramipril
Number analyzed (Participants) | 190 | 190
mm Hg
  Baseline | 72.7 (10.44) | 71.9 (9.85)
  Week 8 | 54.7 (13.87) | 58.9 (13.98)
  Change from baseline to week 8 | -18.0 (12.14) | -13.0 (12.12)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Aliskiren HCTZ | Ramipril
Serious Adverse Events (participants affected / at risk) | 4/193 | 2/193
Other Adverse Events (participants affected / at risk) | 14/193 | 17/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren HCTZ (N=193) | Ramipril (N=193)
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren HCTZ (N=193) | Ramipril (N=193)
Headache (Nervous system disorders) | 14 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.